CLINICAL TRIAL: NCT06862596
Title: A Multicenter, Randomized, Placebo-controlled, Double-blind Clinical Trial: The Efficacy and Safety of Mexiletine Hydrochloride for Amelioration of Motor Dysfunction in Spinal and Bulbar Muscular Atrophy
Brief Title: Clinical Trial of Mexiletine Hydrochloride for Spinal and Bulbar Muscular Atrophy
Acronym: Med-SBMA
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Masahisa Katsuno (Other)
Responsible Party: Sponsor-Investigator, Masahisa Katsuno, Professor, Nagoya University
Organization: Nagoya University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAMCR-026; jRCT2041240174 (Other: Japan Registry of Clinical Trials)
Record Dates: First submitted 2025-02-26; First posted 2025-03-06 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-03

CONDITIONS: Spinal and Bulbar Muscular Atrophy
MeSH Terms: conditions — Bulbo-Spinal Atrophy, X-Linked | interventions — Mexiletine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mexiletine group (Active Comparator)
  Interventions: Drug: Mexiletine hydrochloride
- Placebo group (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Mexiletine hydrochloride — Mexiletine hydrochloride 300 mg is administered orally divided into three times a day after meals for 12 weeks.
  Arms: Mexiletine group
Other: Placebo — Placebo is administered orally divided into three times a day after meals for 12 weeks.
  Arms: Placebo group

SUMMARY:
The purpose of this clinical trial is to evaluate the efficacy and safety of mexiletine hydrochloride in patients with spinal and bulbar muscular atrophy.

The main questions it aims to answer are:

Does mexiletine hydrochloride improve the ALSFRS-R score in spinal and bulbar muscular atrophy patients?

Participants will:

Take mexiletine hydrochloride or a placebo every day for 3 months Visit the hospital once every 4 weeks for evaluations.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients with a CAG repeat count of 38 or more for the androgen receptor gene in genetic testing and a confirmed diagnosis of SBMA
2. Patients with muscle weakness (limb weakness and atrophy, or bulbar palsy) due to lower motor neuron lesion
3. Patients with a total ALSFRS-R score of ≥ 24 and ≤ 42 at screening
4. Patients who are at least 18 years old and less than 80 years old at the time of consent
5. Patients who give their voluntary written consent after having received adequate information on this study (However, if the patient is unable to sign the consent form due to the condition of the disease, a person equivalent to a regal representative must be present to provide written explanation, the prospective candidate must verbally consent to participate in the study, and a person equivalent to a regal representative must sign the consent form on behalf of the patient. The person who is to be the regal representative may sign the document on his/her behalf, noting the circumstances and his/her relationship to the subject.)

Exclusion Criteria:

1. Patients who have participated or are participating in a clinical trial within 12 weeks prior to enrollment
2. Patients with a history of hypersensitivity to any component of this drug product
3. Patients with a conduction disturbance (such as second- or third-degree atrioventricular block without a pacemaker, or left bundle branch block)
4. Patients with Brugada-type ECG
5. Patients with severe heart failure or heart disease (myocardial infarction, valvular disease, cardiomyopathy, etc.)
6. Patients with sinus bradycardia (<50 beats/minute)
7. Patients with systolic blood pressure of 90 mmHg or less
8. Patients with serum potassium level less than 3.5 mmol/L
9. Patients on antiarrhythmic drugs
10. Patients on antiepileptic drugs that affect to sodium channels
11. Patients on theophylline
12. Patients on narcotics
13. Patients who used Mexiletine within 1 month prior to enrollment or used Mexiletine for expectations of improvement in symptoms of SBMA
14. Patients with serious complications
15. Patients who cannot agree to use contraception during the study period
16. Other Patients deemed inappropriate by the investigator or subinvestigator

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) score | at 4weeks
  The ALSFRS-R is a comprehensive severity index comprising 12 items covering bulbar, upper limb, lower limb, and respiratory symptoms to evaluate the ADLs of patients with amyotrophic lateral sclerosis (ALS). Each item is rated on a five-point scale from 0 (worse) to 4 (better), and a total score (miniimum 0point and maximum 48 point) is calculated.

SECONDARY OUTCOMES:
ALSFRS-R Score | up to 12 weeks
  The ALSFRS-R is a comprehensive severity index comprising 12 items covering bulbar, upper limb, lower limb, and respiratory symptoms to evaluate the ADLs of patients with ALS. Each item is rated on a five-point scale from 0 (worse) to 4 (better), and a total score (miniimum 0point and maximum 48 point) is calculated.
Spinal and Bulbar Muscular Atrophy Functional Rating Scale (SBMAFRS) score | up to 12 weeks
  The SBMAFRS is a disease-specific motor function assessment scale for Spinal and Bulbar Muscular Atrophy (SBMA).The SBMAFRS is a comprehensive severity index comprising 14 items covering bulbar, upper limb, lower limb, and respiratory symptoms to evaluate the ADLs of patients. Each item is rated on a five-point scale from 0 (worse) to 4 (better), and a total score (miniimum 0point and maximum 56 point) is calculated.
Grip strength | up to 12 weeks
  Grip strength (kg) is set to evaluate the upper limb motor function of patients with SBMA.
Tongue pressure | up to 12 weeks
  Tongue pressure (kPa) is set to evaluate the bulbar function of patients with SBMA.
Timed walk test (4.6 meters) | up to 12 weeks
  The timed walk test (4.6 meters) is an evaluation index for muscle weakness and atrophy of the lower limbs that measures the walking time (in seconds).
6-minute walk test | up to 12 weeks
  The 6-minute walk test is an evaluation index for lower limb muscle weakness and muscle atrophy that measures the walking distance (in meters).
Respiratory function test (Forced Vital Capacity (FVC)) | up to 12 weeks
  FVC (actual value (L) and predicted rate (%) (%FVC)) is set to evaluate for respiratory function.
Respiratory function test (Peak Expiratory Flow (PEF)) | up to 12 weeks
  PEF (actual value (L/sec) and predicted rate (%) (%PEF)) is set to evaluate for respiratory function.

CONTACTS AND LOCATIONS:
Overall Officials: Masahisa Katsuno, PhD, MD, Principal Investigator — Nagoya University Hospital
Locations (5):
- Japan (5):
  - Tokyo University Hospital, Bunkyō City
  - Chiba University Hospital, Chiba
  - Hokkaido University Hospital, Sapporo
  - Jichi Medical University Hospital, Shimotsuke
  - Osaka University Hospital, Suita

IPD SHARING:
Plan to Share IPD: Yes
If the principal investigator, clinical trial office, main stakeholder conclude that secondary use of individual data obtained in this clinical trial is beneficial for additional analysis, the secondary use of data excluding personal information will be acceptable after publication of results.